CLINICAL TRIAL: NCT04127032
Title: Internet-Delivered Cognitive Behaviour Therapy (ICBT) for Public Safety Personnel (PSP): Examination of Engagement, Outcomes, Strengths and Challenges
Brief Title: Internet-Delivered Cognitive Behaviour Therapy for Public Safety Personnel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Government of Canada (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-157
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Depression, Anxiety; Psychological Trauma
Keywords: Internet; Cognitive Behavioral Therapy; Telemedicine
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tailored ICBT for PSP (Experimental): Therapist-guided, Internet-delivered cognitive behavioral therapy tailored specifically for Canadian public safety personnel.
  Interventions: Behavioral: PSP Wellbeing Course

INTERVENTIONS:
Behavioral: PSP Wellbeing Course — A tailored ICBT intervention will be delivered to public safety personnel who report symptoms of depression, anxiety, or posttraumatic stress. Clients will choose whether they prefer weekly therapist support, twice-weekly support, or monitored optional support. The intervention is designed to be completed in 8 weeks, but clients will be able to extend their access to therapist support by an additional 8 weeks (i.e., up to 16 weeks in total).

SUMMARY:
This study evaluates a transdiagnostic Internet-delivered cognitive behavioural therapy (ICBT) recently tailored for Canadian public safety personnel (PSP) reporting symptoms of depression, anxiety, or posttraumatic stress. Outcomes of interest include engagement with the intervention, changes in symptoms and functioning, and strengths and limitations of implementing ICBT with Canadian PSP.

DETAILED DESCRIPTION:
Background:

Public Safety Personnel (PSP) is a term that broadly encompasses personnel who ensure the safety and security of Canadians across jurisdictions, including, but not necessarily limited to, public safety communications officials (e.g., call centre operators/dispatchers), correctional employees, firefighters, paramedics, border services personnel, operational and intelligence personnel, search and rescue personnel, and police officers. As a function of their vocations, PSP are frequently exposed to traumatic events (e.g., threatened or actual physical assaults, sexual violence, fires, and explosions) and are at risk of post-traumatic stress injuries. Results from a recent survey with a large Canadian PSP sample showed 44.5% screened positive for one or more mental health disorders, which is much higher than the 10.1% diagnostic rate among the Canadian general public. For many Canadian PSP access to in-person evidence-based care is impeded for several reasons, including preference to self-manage symptoms, geographic barriers (e.g., difficulty accessing care while deployed to remote locations), logistical barriers (e.g., shift work limits access to standard service hours), stigma (e.g., perceptions of being evaluated negatively for having mental health concerns), growing waiting-lists, and limited resources (e.g., insufficient access to mental health care coverage).

Transdiagnostic Internet-delivered cognitive behaviour therapy (ICBT) represents a convenient method for PSP to access care for mental health concerns, such as depression, anxiety, and post-traumatic stress. In transdiagnostic ICBT, clients receive access to standardized lessons that provide the same information and skills as traditional face-to-face CBT. Divergent mental health symptoms are targeted within transdiagnostic ICBT by educating clients in strategies that apply to multiple conditions (e.g., cognitive restructuring, graded exposure); this helps to ensure multiple concerns are addressed in an efficient manner. This is important given high rates of mental health comorbidity. In addition to weekly lessons, clients are encouraged to complete homework assignments to facilitate learning. Research shows that transdiagnostic ICBT is effective at reducing symptoms of anxiety, depression and trauma and there is also evidence that the findings of research trials translate into routine clinic settings. Most commonly, ICBT is delivered with brief once weekly e-therapist assistance (~20 minutes) via the telephone or secure email over ~8 weeks. There are also encouraging research results that clients can benefit with lower levels of support, such as when treatment is largely self-directed but with automated reminder emails, e-therapist monitoring and optional e-therapist support as needed by clients.

Research purpose:

The purpose of the current research project is to explore outcomes of a transdiagnostic ICBT course that is specifically tailored for PSP (e.g., case examples are relevant to PSP), referred to as the PSP Wellbeing Course. Of particular interest in this study are: 1) the usage of the PSP Wellbeing Course among PSP who are informed about the PSP Wellbeing Course (e.g., # enrolling, completion rates, use of e-therapist support); 2) outcomes of the PSP Wellbeing Course with respect to diverse outcome measures (e.g., depression, anxiety, trauma, functioning) measured at 8, and 26 week follow-up; and 3) strengths and challenges of the PSP Wellbeing Course when offered to Canadian PSP. In order to take part, PSP will first complete an online questionnaire and telephone screening to assess whether they meet the following inclusion criteria: 1) 18 years of age or older; 2) resident of the Canadian provinces of Saskatchewan, Quebec, Nova Scotia, New Brunswick, Prince Edward Island or Ontario; 3) not endorsing high suicide risk or recent suicide attempts in the past year; 4) able to access and comfortable using computers and the internet; 5) not seeking help primarily for alcohol and or drugs, bipolar disorder, or psychotic symptoms; and 6) willing to provide an emergency contact unless the participant does not have a physician and the clinician assesses the need for an emergency contact as low during the telephone screening. The PSP Wellbeing Course will be delivered by trained providers with graduate training in psychology or social work or graduate students under supervision. Of note, the program was first offered in Saskatchewan and later translated to French and offered to PSP who reside in Quebec as well (update: recruitment in Quebec began on September 23, 2020). The program was also expanded to PSP in Nova Scotia, New Brunswick, and Prince Edward Island in February 2022, as well as to PSP in Ontario in March 2023. Of note, a purely self-guided version of the PSP Wellbeing Course (i.e., without therapist guidance) was made available to PSP anywhere in Canada in English on December 1st, 2021 and in French on November 19th, 2022. The primary research questions to be answered include:

1. ENGAGEMENT: How many PSP will enroll in and complete the PSP Wellbeing Course? What will be the uptake of optional e-therapist support, versus 1x week or 2x week e-therapist support? What will be the length of support selected (8 week-16 week)?
2. OUTCOMES: What will be the impact of the PSP Wellbeing Course on symptom improvement and functioning at 8, 26, and 52 weeks post-enrollment? What factors will predict outcomes (e.g., symptom severity, demographics, engagement)? Please note: as of December 2024, we are exploring the impact of the PSP Wellbeing Course on symptom improvement and functioning at 8, and 26 weeks post-enrollment. The impact of this course at weeks 8, 26, and 52 was previously explored and has been published
3. IMPLEMENTATION: What are stakeholder experiences, positive and negative, with the PSP Wellbeing Course? What are the suggested improvements to ICBT to meet the needs of PSP?

Significance:

This project will provide information that will inform future use of ICBT to assist PSP with common mental health concerns. Data will be extracted and analyzed on a quarterly basis in order to provide a preliminary evaluation of engagement, outcomes and implementation experiences and determine if adjustments to ICBT are required. Once adjustments are completed or deemed unnecessary, data will be extracted and analyzed biannually.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* residing in a Canadian province or territory in which PSPNET is able to offer services
* endorsing symptoms of anxiety, depression, or post-traumatic stress
* able to access a computer and internet service
* willing to provide a physician as emergency contact unless the participant does not have a physician and the clinician conducting the telephone screening assesses the need for an emergency contact to be low.

Exclusion Criteria:

* high suicide risk
* suicide attempt or hospitalization in the last year
* primary problems with psychosis, alcohol or drug problems, mania
* currently receiving regular psychological treatment for anxiety or depression
* not present in Canada during treatment
* concerns about ICBT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in depression | screening and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 26, and 52 weeks (note: as of December 2024, we are no longer collecting data at 52 weeks).
  Patient Health Questionnaire - 9 Item (PHQ-9). Higher total scores indicate greater severity of depression. Scores range from 0 to 27. Note: this measure is only administered at weeks 9 through 16 for clients who are still engaged in treatment at those timepoints.
Change in anxiety | screening and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11,12, 13, 14, 15, 16, 26, and 52 weeks (note: as of December 2024, we are no longer collecting data at 52 weeks).
  Generalized Anxiety Disorder - 7 Item (GAD-7). Higher total scores indicate greater severity of anxiety. Scores range from 0 to 21. Note: this measure is only administered at weeks 9 through 16 for clients who are still engaged in treatment at those timepoints.
Change in posttraumatic stress | screening and 8, 26, and 52 weeks (note: as of December 2024, we are no longer collecting data at 52 weeks).
  PTSD Checklist for DSM-5 (PCL-5). Higher total scores indicate greater severity of posttraumatic stress. Scores range from 0 to 80.
Change in posttraumatic stress | 1, 2, 3, 4, 5, 6, 7, 9, 10, 11, 12, 13, 14, 15 and 16 weeks
  Abbreviated PTSD Checklist - Civilian Version (PCL-C). Higher total scores indicate greater severity of posttraumatic stress. Scores range from 5 to 30. Note: this measure is only administered at weeks 9 through 16 for clients who are still engaged in treatment at those timepoints.

SECONDARY OUTCOMES:
Change in panic symptoms | screening and 8, 26, and 52 weeks (note: as of December 2024, we are no longer collecting data at 52 weeks).
  Panic Disorder Severity Scale-Self Report (PDSS-SR), 2-item version. Higher total scores indicate greater severity of panic symptoms. Scores range from 0 to 8. Note: this measure replaced the full PDSS-SR on October 6, 2023.
Change in social anxiety | screening and 8, 26, and 52 weeks (note: as of December 2024, we are no longer collecting data at 52 weeks).
  Mini-Social Phobia Inventory (Mini-SPIN): Higher total scores indicate greater severity of social anxiety, with scores ranging from 0 to 12. In the English version of the course, the Mini-SPIN replaced the 6-item Social Interaction Anxiety Scale (SIAS-6) and the 6-item Social Phobia Scale (SPS-6) on October 6th, 2023. In the French version of the course, it replaced the Social Interaction Phobia Scale (SIPS) on March 20th, 2024.
Change in anger | screening and 8, 26, and 52 weeks (note: as of December 2024, we are no longer collecting data at 52 weeks).
  Dimensions of Anger Reactions (DAR-5) scale. Higher total scores indicate greater severity of anger problems. Scores range from 0 to 20.
Change in sleep problems | screening and 8, 26, and 52 weeks (note: as of December 2024, we are no longer collecting data at 52 weeks).
  Insomnia Severity Index (ISI). Higher total scores indicate greater severity of sleep problems. Scores range from 0 to 28. Note: this measure was added on December 3, 2020.
Other sleep problems | screening
  SLEEP-50 Questionnaire. This questionnaire consists of 50 items spanning 9 subscales. However, instead of administering and scoring the entire questionnaire, we are administering only 21 items for descriptive purposes. Note: this measure was added on December 3, 2020.
Alcohol use | screening
  Alcohol Use Disorders Identification Test (AUDIT). Higher scores indicate greater alcohol consumption and alcohol-related problems. Scores ranger from 0 to 40.
Drug use | screening
  Drug Use Disorders Identification Test-C (DUDIT-C). Higher scores indicate greater drug use and drug-related problems. Scores ranger from 0 to 16. Note: this measure replaced the full DUDIT in December 2024.
Change in functioning | screening and 4, 8, 12, 26, and 52 weeks (note: as of December 2024, we are no longer collecting data at 52 weeks).
  Work and Social Adjustment Scale (WSAS). Higher total scores indicate a greater degree of impairment. Total scores range from 0 to 40. Note: this measure is only administered at 12 weeks for clients who are still engaged in treatment at this timepoint. Note: this measure replaced the Sheehan Disability Scale (SDS).
Change in resiliency | screening and 8, 26, and 52 weeks (note: as of December 2024, we are no longer collecting data at 52 weeks).
  Brief Resiliency Scale (BRS). Higher total scores indicate greater resiliency. Total scores represent mean scores across the six items of the scale and range from 0 to 5. Note: this measure was added on December 3, 2020.
Change in use of health services | screening and 8, 26, and 52 weeks (note: as of December 2024, we are no longer collecting data at 52 weeks).
  Health Service Use Questionnaire is a bespoke questionnaire that assesses the use of health services for mental health problems.
Treatment satisfaction | week 8
  Treatment Satisfaction Questionnaire. A bespoke questionnaire consisting of 32 items with varying response formats measuring treatment satisfaction and perceived treatment credibility. Items are not designed to be combined into a unitary measure.
Working alliance | week 8
  Working Alliance Inventory - Short Revised (WAI-SR). Higher scores indicate greater working alliance. Scores in three distinct domains of working alliance each range from 4 to 20.
Lifetime Traumatic Events History | screening and 52 weeks (note: as of December 2024, we are no longer collecting data at 52 weeks).
  Life Events Checklist for DSM-5 (LEC-5). A checklist of common traumatic events used to establish the nature of the traumatic events a respondent has experienced. This questionnaire is not intended to be scored.
Worst Traumatic Event | screening and 52 weeks (note: as of December 2024, we are no longer collecting data at 52 weeks).
  Worst Traumatic Event Questionnaire. A checklist of common traumatic events used to establish the nature of the single worst traumatic event a respondent has experienced. This questionnaire is not intended to be scored.
Engagement and Homework Compliance | 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 weeks
  Homework Reflection. A bespoke questionnaire consisting of 8 items with varying response formats, designed to measure engagement with treatment tasks and help alert therapists to any challenges clients face. Items are not designed to be combined into a unitary measure. Note: this measure is only administered at 9, 10, 11, and 12 weeks for clients who are still engaged in treatment at those timepoints.
Change in Moral Injury | screening, 8 and 26 weeks.
  Moral Injury Outcome Scale - Abbreviated Winter Campaign version. High total scores indicate greater levels of current moral injury. Scores range from 0 - 56. Note: this measure was added in December 2024

CONTACTS AND LOCATIONS:
Overall Officials: Heather D Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- Department of Psychology and Canadian Institute for Public Safety Research and Treatment, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Price JA, McCall HC, Demyen SA, Spencer SM, Katz BM, Clairmont AP, Hadjistavropoulos HD. Optimization of Internet-Delivered Cognitive Behavioral Therapy for Canadian Leaders Within Public Safety: Qualitative Study. J Med Internet Res. 2025 Apr 17;27:e72321. doi: 10.2196/72321. PMID 40245389
- [Derived] Price JA, Gregory J, McCall HC, Landry CA, Beahm JD, Hadjistavropoulos HD. Client Perspectives of Case Stories in Internet-Delivered Cognitive Behavioral Therapy for Public Safety Personnel: Mixed Methods Study. JMIR Form Res. 2024 Oct 25;8:e64454. doi: 10.2196/64454. PMID 39453705
- [Derived] Hadjistavropoulos HD, McCall HC, Thiessen DL, Huang Z, Carleton RN, Dear BF, Titov N. Initial Outcomes of Transdiagnostic Internet-Delivered Cognitive Behavioral Therapy Tailored to Public Safety Personnel: Longitudinal Observational Study. J Med Internet Res. 2021 May 5;23(5):e27610. doi: 10.2196/27610. PMID 33949959
- See also: Additional information about the PSP Wellbeing Course. — https://www.pspnet.ca/en/for-psp/online-courses/therapist-guided-psp-wellbeing-course